CLINICAL TRIAL: NCT05365724
Title: A Study to Evaluate the Safety and Immunogenicity of Omicron COVID-19 Vaccine (Vero Cell), Inactivated in Population 18 Years Old of Age and Above With no Vaccination History of COVID-19 Vaccine
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Omicron COVID-19 Vaccine (Vero Cell), Inactivated in Population 18 Years Old of Age and Above
Acronym: COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry); Shulan (Hangzhou) Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNBG-BIBP-O-2022003
Record Dates: First submitted 2022-04-30; First posted 2022-05-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: COVID-19; Omicron; inactivated vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subjects aged 18-59 years old (Experimental)
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated
- subjects aged 60 years old and above (Experimental)
  Interventions: Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: Omicron COVID-19 Vaccine (Vero Cell), Inactivated — 2 doses of vaccine according to the immunization schedule of 0, 21-28 days

SUMMARY:
This is a non-randomized, open-label, externally controlled study to evaluate the safety and immnunogenicity of the Omicron COVID-19 Vaccine (Vero Cell), Inactivated in population aged 18 years old and above with no vaccination history of the COVID-19 vaccine. 200 health subjects will be recruited in this study, including 150 aged 18-59 years old and 50 aged 60 years old and above. All subjects will be received 2 doses of Omicron COVID-19 Vaccine (Vero Cell), Inactivated according to the immunization schedule of 0, 21-28 days. The change in neutralizing antibody level at 28 days after the second dose was used to determine whether to receive a further booster dose for ≥3 months.

The occurrence of adverse events within 28 days and serious adverse events within 6 months after vaccination will be observed. In addition, blood samples will be collected on Day 0 before vaccination,Day 14 after dose 1, before dose 2 and on day 14, 28 and month 3, 6, 9, 12 after dose 2. Serum antibody levels, cellular immune responses will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 years old and above.
* By asking for medical history and physical examination, the investigator judged - that the health condition is well.
* Female subjects of childbearing age are not nursing or pregnant at the time of enrolment (negative urine pregnancy test) and have no family planning within the first 12 months after enrolment. Effective contraceptive measures have been taken within 2 weeks before inclusion.
* During the whole follow-up period of the study, be able and willing to complete the whole prescribed study plan.
* With self-ability to understand the study procedures, the informed consent & voluntarily sign an informed consent form and be able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

* Confirmed or suspected cases of SARS-CoV-2 Infection.
* Has a history of SARS, MERS, SARS-CoV-2 infection (self-report, on-site inquiry).
* Has received COVID-19 vaccine (include mRNA, recombinant protein vaccines, vector vaccines, inactivated vaccines, etc.)
* Axillary body temperature > 37.3 ℃ before vaccination
* Previous severe allergic reactions to vaccination (such as acute allergic reactions, urticaria, dyspnea, angioneurotic edema or abdominal pain) or allergy to known ingredients of inactivated SARS-CoV-2 vaccine have occurred (self-report, on-site inquiry).
* History of hospital-diagnosed thrombocytopenia or other coagulation disorder
* Known immunological impairment or low level with hospital diagnosis
* History of uncontrolled epilepsy, other progressive neurological disorders, or Guillain-Barre syndrome (self-report, on-site inquiry).
* Known or suspected concomitant serious diseases include: respiratory disease, acute infection or active chronic disease, liver and kidney disease, severe diabetes, malignant tumor, infection or allergic skin disease, HIV infection.
* Severe cardiovascular disease (cardiopulmonary failure, uncontrolled hypertension, etc.) diagnosed by the hospital, active chronic respiratory disease
* Live attenuated vaccine is inoculated within 1 month before this vaccination
* other vaccines are inoculated within 14 days before this vaccination.
* be participating in or plan to participate in other vaccine clinical trials during this study.
* Contraindications related to vaccination as considered by other investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
The Geometric Mean Titer (GMT) of neutralizing antibody against Omicron SARS-CoV-2 | On Day 28 after Dose 2
The four-fold increase rate of neutralizing antibody against Omicron SARS-CoV-2 | On Day 28 after Dose 2
Incidence of adverse reactions | within 28 days after vaccination

SECONDARY OUTCOMES:
The Geometric Mean Titer (GMT) of neutralizing antibody against Omicron SARS-CoV-2 | On Day 14 after Dose 2
The four-fold increase rate of neutralizing antibody against Omicron SARS-CoV-2 | On Day 14 after Dose 2
The incidence of any adverse reactions/events | 28 days after each immunization
The incidence of serious adverse events (SAE) and adverse events special interest (AESI) | From the beginning of the first dose to 12 months after the second immunization
The neutralizing antibody GMT | on 3rd month, 6th month, 9th month, and 12th month after Dose 2
The proportion of subjects of neutralizing antibody GMT ≥1:16，≥1:32 and ≥1:64 | on 3rd month, 6th month, 9th month, and 12th month after Dose 2

OTHER OUTCOMES:
The neutralizing antibody GMT to different variants of SARS-CoV-2 | On Day 28 after Dose 2
The IgG antibody lever against Omicron SARS-CoV-2 | On Day 14 and 28 after Dose 2
The incidence of COVID-19 cases | From 14 day after Dose 2
The incidence of severe cases of COVID-19, including deaths accompanied by COVID-19) | From 14 day after Dose 2

CONTACTS AND LOCATIONS:
Overall Officials: Lanjuan Li, Principal Investigator — Shulan (Hangzhou) Hospital
Locations (1):
- Shulan (hangzhou) Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No